CLINICAL TRIAL: NCT06502821
Title: Preferences of Israeli New Physiotherapists in Choosing Their Future Workplace
Status: Recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PHD, Prof., University of Haifa
Other Study IDs: 433/23
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Workplace

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- students: 4th year students of physical therapy
  Interventions: Other: questtionnaire
- young physiotherapists: physiotherapists 1-3 years in the profession
  Interventions: Other: questtionnaire
- experienced physical therapist: physical therapists with over 10 years in profession
  Interventions: Other: questtionnaire

INTERVENTIONS:
Other: questtionnaire — questionnaire regarding workplace preferences and the factors influencing choosing a career in physiotherapy

SUMMARY:
This study aim to create a multidimensional body of knowledge on the factors influencing physiotherapy graduates in Israel in choosing a workplace, satisfaction with the chosen framework, and intergenerational differences in these factors. In addition, to examine the relationship between the factors for choosing a professional career in physiotherapy and choosing a workplace

DETAILED DESCRIPTION:
The study will be mixed methods and will include: focus groups for the accuracy of the content of the questionnaires (5 students, 5 physiotherapists), a preliminary study to examine the clarity and understanding of the questionnaires (10 students,20 physiotherapists), and a cross-sectional study using online questionnaires to examine workplace preferences and the factors influencing choosing a career in physiotherapy among fourth-year students, young physiotherapists and experienced physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* physiotherapists

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: students for physical therapy, during their 4th year of studying, and experienced physical therapists
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
choosing a profession | baseline
  Rating reasons for choosing physical therapy as a profession. questionnaire with 16 statements, each statement will be evaluated on a scale from 1(not at all) to 4 (very much)
choosing workplace | baseline
  Rating reasons for choosing workplace. questionnaire with 22 statements, each statement will be evaluated on a scale from 1(not at all) to 4 (very much)

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided